CLINICAL TRIAL: NCT07150689
Title: Assessment of Outcome of Bronchoscopy in Pediatric Patients With Suspected Foreign Body Aspiration Attending at Assiut University Children Hospital
Brief Title: Outcome of Bronchoscopy in FB Aspiration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marsail Refat Kadry, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FB bronchoscopy
Record Dates: First submitted 2025-08-08; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-07

CONDITIONS: Foreign Body Aspiration
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Masking Description: Masking Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Rigid Bronchoscopy (Active Comparator): Standard of care in most pediatric centers; performed under general anesthesia to visualize and remove FB. Gold standard for both diagnosis and treatment
  Interventions: Procedure: Rigid bronchoscopy
- Flexible Bronchoscop (Experimental): Flexible scope used for diagnosis and sometimes removal (especially in distal airways or when FB is small). Evaluate if less invasive flexible bronchoscopy can be effective.
  Interventions: Procedure: Flexible scope
- Combined Approach (Experimental): Initial flexible bronchoscopy for diagnosis and airway inspection, followed by rigid bronchoscopy for removal if needed. Compare efficiency and safety of combined method.
  Interventions: Procedure: Combined Flexible-Rigid Bronchoscopy
- Imaging-Guided Approach (Experimental): High-resolution CT or virtual bronchoscopy first; bronchoscopy only if imaging suggests FB. Assess if imaging can reduce unnecessary bronchoscopies.
  Interventions: Procedure: Imaging-Guided Bronchoscopy

INTERVENTIONS:
Procedure: Rigid bronchoscopy — Participants will undergo rigid bronchoscopy under general anesthesia using an age-appropriate rigid bronchoscope. The airway will be systematically inspected. Any identified foreign body will be removed using appropriate retrieval devices (optical forceps, retrieval basket, suction). Post-removal, the airway will be re-examined to confirm clearance and detect trauma.
  Arms: Rigid Bronchoscopy
Procedure: Flexible scope — Participants will undergo flexible fiberoptic bronchoscopy under sedation or general anesthesia. The bronchoscope will be inserted transorally or transnasally. The airway will be inspected, and foreign body retrieval attempted using retrieval baskets, forceps, or cryoprobe
  Arms: Flexible Bronchoscop
Procedure: Combined Flexible-Rigid Bronchoscopy — Initial flexible bronchoscopy will be performed to locate the foreign body and inspect distal airways, followed by rigid bronchoscopy for definitive removal.
  Arms: Combined Approach
Procedure: Imaging-Guided Bronchoscopy — Participants will undergo pre-procedure high-resolution CT or virtual bronchoscopy. Based on imaging, either rigid or flexible bronchoscopy will be performed, targeting the suspected location to reduce procedure time.
  Arms: Imaging-Guided Approach

SUMMARY:
Outcome of Bronchoscopy in Pediatric patient with foreign body aspiration

ELIGIBILITY:
Inclusion Criteria:

* children less than 18 years with suspected foreign body aspiration

Exclusion Criteria:

* children with congenital airway anomalies other than foreign body aspiration

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Rate of Successful Foreign Body Removal | During bronchoscopy procedure (intra-operative, within 24 hours of intervention).
  The proportion of patients in whom the foreign body is completely removed during the initial bronchoscopy procedure, as confirmed by direct visualization and/or post-procedure imaging.

SECONDARY OUTCOMES:
Incidence of procedure-related complications (within 24 hours). | Intra-procedure and up to 24 hours post-procedure.
  Number of patients who experience complications such as hypoxia (SpO₂ < 90%), bleeding, airway trauma, pneumothorax, or cardiac arrhythmia.